CLINICAL TRIAL: NCT00704756
Title: An Observational Multi-Center Study Exploring the Association of Safety, Patient Characteristics, Virological, and Histological Parameters With Patient Outcome (Relapse Rate, Achievement of Sustained Viral Response in Daily Clinical Practice in Belgium- PEGIMPACT
Brief Title: An Observational Study of Patients With Chronic Hepatitis C Undergoing Treatment With PegIntron and Rebetol in Clinical Practice in Belgium (Study P05494)(WITHDRAWN)
Acronym: PEGIMPACT
Status: Withdrawn | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05494
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Patients with chronic hepatitis C treated with PegIntron and Rebetol in clinical practice in Belgium.
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — PegIntron administered at 1.5 μg/kg body weight/week subcutaneously for up to 24 wks (Genotype [G] 2,3/low viral load G 1) or 48 weeks for (G 1,4,5)
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered based on body weight 800-1200 mg/day (<65 kg : 800 mg, 65 - 85 kg : 1000 mg, >85 kg : 1200 mg) orally for up to 24 wks (Genotype [G] 2,3/low viral load G 1) or 48 weeks for (G 1,4,5)
  Other Names: SCH 18908

SUMMARY:
This is an observational study of patients undergoing treatment with PegIntron and Rebetol for chronic hepatitis C in clinical practice in Belgium. Treatment will not be administered as part of the study. Safety parameters will be assessed retrospectively. Efficacy parameters, such as relapse rates and sustained virologic response rates, will be assessed prospectively. The objective of the study is to examine any associations between safety, virologic, histologic, demographic parameters and patient outcome (relapse rates and sustained virologic response rates).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult (18 years or older) subjects for whom the treating physician has decided to start treatment with PegIntron® and Rebetol® and reaching the End-of-Treatment time point.
* For the prospective component, evidence of treatment response at EOT after a complete course of therapy as per SmPC.
* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be diagnosed with chronic hepatitis C (genotypes 1, 2, 3, 4, 5 or 6).
* Subjects must be free of any clinically significant disease that would interfere with study participation.

Exclusion Criteria:

* For prospective component of the study: patients not achieving End-of-Treatment response after a complete course of therapy as per SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C treated with PegIntron and Rebetol in clinical practice in Belgium.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Safety parameters: common adverse events [AEs], drug-to-drug interaction AEs, and dose modifications | Assessed retrospectively in patients treated for up to 24 wks (Genotype [G] 2,3/low viral load G 1) or 48 weeks for (G 1,4,5) and reaching End-of-Treatment.

SECONDARY OUTCOMES:
Relapse rates and Sustained Virologic Response (SVR) rates and their association with demographic, virologic, histological, and safety parameters | Assessed prospectively at End-of-Treatment (EOT) and 24 weeks post-treatment
Predictors of response at End-of-Treatment | Assessed at the End-of-Treatment

REFERENCES:
- [Result] Van Vlierberghe H, Adler M, Bastens B, Colle I, Delwaide J, Henrion J, Horsmans Y, Michielsen P, Golstein P, Mulkay JP, Van Steenbergen W, Yap P, Nevens F, Denys AM, Brasseur JP. Effectiveness and tolerability of pegylated interferon alfa-2b in combination with ribavirin for treatment of chronic hepatitis C: the PegIntrust study. Acta Gastroenterol Belg. 2010 Jan-Mar;73(1):5-11. PMID 20458844